CLINICAL TRIAL: NCT04631224
Title: Longitudinal Analysis of Oral Communication in Friedreich's Ataxia
Acronym: ORFA
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011-000389-32
Record Dates: First submitted 2020-07-31; First posted 2020-11-17 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2015-08

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Friedreich Ataxia (FA) is a hereditary neurological disease that is associated with a cerebellar syndrome and pyramidal symptoms. Clinical expression varies from one individual to another and throughout the evolution of the disease and is partially related to an abnormal expansion of the GAA triplet repeat in the frataxin gene. Dysarthria, a disorder in the motor production of speech, is always present in the clinical presentation of the disease (Schöls et al. 1997 ; Harding 1981 ; Dürr et al. 1996 ; Delatycki et al. 1999). It has been the subject of specific studies exploring the link between the evolution of dysarthria and disease progression (J. Folker et al. 2010; J. E. Folker et al. 2012; Rosen et al. 2012; Brendel et al. 2013). These studies allowed for the identification of markers for speech disintegration, specific to FA dysarthria, using perceptive voice measures, but also acoustics and objectives for qualifying voice and speech at the same time. The challenge is in finding measures sufficiently appropriate and sensitive to detect the evolution of these indicators throughout the course of the disease (Rosen et al. 2012). The neurological scales that take in to account all signs of a cerebellar syndrome are not sufficiently sensitive (Marelli et al. 2012). In addition, hearing difficulties develop during the course of the disease in addition to visual disturbances (gaze instability) which hinder communication. The ORFA study aims to evaluate oral communication in FA patients and identify appropriate measures that allow for the comparison of dysarthria pre and post-treatment in a clinical trial and can be used for the evaluation of efficacy.

DETAILED DESCRIPTION:
The ORFA research study will depend partly on the EFACTS consortium (European Friedreich's Ataxia Consortium for Translational Studies) in which the French center ICM participates since 2011 (principal investigator Pr Alexandra Durr). The clinical registry EFACTS has included 604 FA patients to date who are followed annually with the goal of collecting clinical and biological information via a database. In Paris, 50 FA patients are followed and receive a complete evaluation at each visit: clinical evaluations, blood test, cardiac evaluation, and neuropsychological evaluation. In addition, ORFA will be closely linked with the CERMOI project, entitled "Integrated functional evaluation of the cerebellum" which will study visual motor disturbances in FA. This project received funding in 2014 through the IHU-A-ICM, Institute of translational and neuroscientific research which includes 4 research teams at the ICM. CERMOI will combine clinical examination, recording of ocular movements, vestibular testing, gait and posture tests.

ORFA will enable to assess the difficulties in articulation and hearing in FA patients and correlate this data with clinical and biological data collected in EFACTS. 50 francophone FA patients will be followed for 2 visits with a one-year interval in between.

ELIGIBILITY:
Inclusion Criteria:

* To have Friedreich's Ataxia.
* To be francophone
* Being a reader
* Agreeing to be part of a research protocol and longitudinal follow-up
* Agree to provide access to medical records

Exclusion Criteria:

* Non-French speaking
* Psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * To have Friedreich's Ataxia.
  * To be francophone
  * Being a reader
  * Agreeing to be part of a research protocol and longitudinal follow-up
  * Agree to provide access to medical records
  Exclusion Criteria:
  * Non-French speaking
  * Psychiatric disorders
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
To identify a sensitive marker of disease progression in Friedreich's Ataxia patients by assessing the speech, voice, oromotor function, and hearing. | Longitudinal timeframe with a first evaluation at baseline and second evaluation one year later
  - Speech therapy assessment: We conduct a statistical study to cross-reference independent variables (age, sex…) and dependent variables. This is to identify relevant and sensitive metrics to capture changes over one year. Dysarthria is assessed by the compensations implemented by patients to maintain the intelligibility of their speech. For example, patients can compensate for their difficulty by slowing the speech flow to maintain good intelligibility. Speech therapy is based on the understanding of these compensation phenomena and uses them in rehabilitation.
  - Recording of the hearing: This non-invasive examination will include tonal audiometry: detection of perception thresholds for sounds of different frequencies and voice audiometry to assess comprehension and intelligibility. This assessment may be supplemented by studying nerve conduction along the auditory pathways. These examinations help to identify the modalities of hearing rehabilitation.